CLINICAL TRIAL: NCT00357344
Title: Weight Changes and the Brain (Study of the Effects of a Large and Intentional Weight Loss Induced by Roux-en-Y Gastric Bypass on Brain Tissue Composition of Obese Patients Using Magnetic Resonance Imaging and Voxel-Based Morphometry)
Brief Title: Study of Effects From Gastric Bypass Weight Loss on Brain Tissue
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906173; 06-DK-N173
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-10-03

CONDITIONS: Weight Loss
Keywords: Obesity; Gray Matter; Eating Behavior; Brain MRI; Body Weight Regulation
MeSH Terms: conditions — Weight Loss; Obesity; Feeding Behavior

SUMMARY:
This study will evaluate how large, intentional weight reduction affects the human brain and possible ways to reverse the changes associated with excess body weight. Subtle changes in some brain regions occur in people who are overweight. Such changes may involve the regulation of eating behavior, though it is not clear whether the changes were present before weight gain or are a consequence. Magnetic resonance imaging (MRI) will be used to study local structures of the brain.

Patients ages 18 to 45 who are undergoing gastric bypass surgery and who are not pregnant or breastfeeding may be eligible for this study. A study group of lean participants will serve as controls. Patients will visit the Phoenix Indian Medical Center for about 3 days at a time for tests. They will have a medical examination, electrocardiogram, and tests of blood and urine. Questionnaires they will complete involve patients' moods and possible influence on eating behaviors, as well as food preferences. A taste test, smell test, and assessment of decision-making processes will be conducted. An oral glucose tolerance test involves a needle placed intravenously (IV) in the arm, for drawing blood after patients drink a sugar solution. The test takes about 3-1/2 hours, with six blood samples taken (about 2 tablespoons total). A meal test also includes use of an IV line. After patients consume a liquid meal, blood will be collected to analyze levels of blood sugar and hormones. For the DEXA scan, which measures body composition, patients will lie still while low-dose X-rays are used for 5 to 10 minutes. Urine will be collected for 1 whole day, to measure cortisol, a hormone. The MRI scan uses a strong magnetic field to obtain images of body organs and tissues. Patients having any metal in the body that may interfere with the scanning machine should not have this test. For the MRI procedure, patients will lie on a table that slides into the enclosed tunnel of the scanner and be asked to lie still. Patients will be able to communicate with the MRI staff at all times during the scan, and they may ask to be removed from the machine at any time.

DETAILED DESCRIPTION:
BACKGROUND: We have identified subtle changes in some brain regions of obese subjects by using a new computerized technique (voxel-based morphometry, VBM) which allows for studying the local structure of the brain by taking very detailed pictures of the brain through magnetic resonance imaging (MRI) and then processing these images with sophisticated statistical software. Some of these regions may interfere with an obese person's ability to predict future consequences of his or her eating behaviors. These changes may explain why people have difficulty losing weight. However, it is not clear whether these changes in the brain are present before or are a consequence of weight gain.

OBJECTIVES: The main aim of this study will be to evaluate the effects of a large and intentional weight reduction on the brains of obese individuals for assessing the possible reversal of the changes associated with excess body weight. Additional objectives will be a) to determine the possible behavioral correlates of the changes in brain tissue composition associated with a large and intentional weight reduction and b) to confirm the results of our previous exploratory analysis showing that human obesity is associated with changes in brain structure in areas related to the regulation of eating behavior.

DESIGN: This is a longitudinal protocol mainly focused on obese patients undergoing roux-en-Y gastric bypass (RYGBP), which represents the most effective approach currently available to achieving substantial weight loss, thus maximizing our chances of detecting significant changes in brain tissue composition. Therefore, we propose to study brain morphology and the metabolic and behavioral characteristics of 40 obese patients undergoing RYGBP prior to and 3, 6, 12, 24, and 48 months after the surgery. Forty lean subjects (at 0, 12, 24, and 48 months) will also be studied for comparison.

OUTCOME MEASURES: The volumes of the different components of the brain by VBM of MRI pictures; metabolic parameters relevant to the relationship between obesity and the brain by measuring fasting concentrations and postprandial responses of some metabolites; the ability to regulate reward and behavior by specific tasks and questionnaires; the ability to detect and discriminate smells by olfaction tests.

ELIGIBILITY:
* INCLUSION CRITERIA

Ethnicity: Caucasian, due to the cross-sectional analysis, upon which the present longitudinal study is based, being made up of Caucasian subjects and the lack of normative data in other racial and ethnic groups

Age 18-45 years, to minimize the confounding role of the well-known effects of aging on brain tissue composition. There is, in fact, compelling evidence from post mortem and in vivo studies that the brain shrinks with age. Neuropathological and CT and MRI morphometric studies indicated that aging predominantly and substantially affects the GM. In addition, deep WM lesions are seen on MRIs in approximately one-third of asymptomatic elderly subjects. Blood pressure also rises with increasing age and can affect brain morphology. Several studies provided evidence of specific patterns in the structural brain correlates of aging, not only globally, between GM and WM compartments, but also locally, within regions of the brain. Therefore, to limit the confounding effect of aging on brain tissue composition, which could theoretically overlap with and confound those of weight loss, the age limit for entering the study will be 45 years.

BMI greater than or equal to 35 kg/m(2) for group 1 and less than 25 kg/m(2) for group 2.

Weight less than or equal to 150 kg (maximum weight allowed on the MRI scanning tables by the manufacturers).

EXCLUSION CRITERIA

History or clinical manifestation of:

* Current smoking
* Type 2 diabetes (according to the World Health Organization diagnostic criteria (63))
* Endocrine disorders, such as Cushing's disease, pituitary disorders, and hypo- and hyperthyroidism
* Pulmonary disorders, including chronic obstructive pulmonary disease that would limit ability to follow the protocol (investigator judgment) and obstructive sleep apnea syndrome; only subjects with mild or exercise-induced asthma on no medications or on beta-adrenergic agonists only (such as albuterol) will be allowed to enter the study
* Cardiovascular diseases, including coronary heart disease, heart failure, arrhythmias, and peripheral artery disease
* Hypertension, as diagnosed and treated by an outside physician or by sitting blood pressure measurement, using an appropriate cuff, higher than 140/90 mmHg on two or more occasions
* Gastrointestinal disease, including inflammatory bowel diseases (e.g. Crohn's disease and ulcerative colitis), malabsorption syndromes (e.g. celiac disease), gastric ulcer (active); only subjects with gastro-esophageal reflux will be allowed to enter the study
* Liver disease, including cirrhosis, active hepatitis B or C, and AST or ALT greater than or equal to 3x normal
* Renal disease, as defined by serum creatinine concentrations greater than or equal to 1.5 mg/dl and/or proteinuria greater than 300 mg/day (200 microgram/min)
* Central nervous system disease, including previous history of cerebrovascular accidents, dementia, and neurodegenerative disorders
* Cancer requiring treatment in the past five years, except for non-melanoma skin cancers or cancers that have clearly been cured or in the opinion of the investigator carry an excellent prognosis (e.g., Stage 1 cervical cancer)
* Conditions not specifically mentioned above may serve as criteria for exclusion at the discretion of the investigators

Personal and/or family history of major psychiatric disorders based upon the DSM-IV (64), including depression, schizophrenia, and psychosis, which may affect brain tissue composition independent of obesity.

Medications acting on the central nervous system and steroidal drugs within 2 months of the baseline study. Non-steroidal anti-inflammatory drugs (NSAID), proton pump inhibitors, and anti-acids will be allowed but discontinued 3 or more days before the admission.

Alcohol and/or drug abuse (more than 3 drinks per day and use of drugs, such as amphetamines, cocaine, heroin, or marijuana).

Contra-indications for MRI, including pacemakers and/or ferromagnetic implants and claustrophobia.

Pregnancy or lactation.

All subjects will be fully informed of the aim, nature, and risks of the study prior to giving written informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80
Dates: Start 2006-05-24; Study Completion 2008-10-03

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - NIDDK, Phoenix, Phoenix, Arizona
  - Good Samaritan Regional Medical Center, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona

REFERENCES:
- [Background] Flegal KM, Carroll MD, Ogden CL, Johnson CL. Prevalence and trends in obesity among US adults, 1999-2000. JAMA. 2002 Oct 9;288(14):1723-7. doi: 10.1001/jama.288.14.1723. PMID 12365955
- [Background] Gustafson D, Rothenberg E, Blennow K, Steen B, Skoog I. An 18-year follow-up of overweight and risk of Alzheimer disease. Arch Intern Med. 2003 Jul 14;163(13):1524-8. doi: 10.1001/archinte.163.13.1524. PMID 12860573
- [Background] Gustafson D, Lissner L, Bengtsson C, Bjorkelund C, Skoog I. A 24-year follow-up of body mass index and cerebral atrophy. Neurology. 2004 Nov 23;63(10):1876-81. doi: 10.1212/01.wnl.0000141850.47773.5f. PMID 15557505